CLINICAL TRIAL: NCT00277667
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Quetiapine Monotherapy in Ambulatory Bipolar Spectrum Disorder With Moderate-to-Severe Hypomanic Symptoms or Mild Manic Symptoms
Brief Title: Study of Quetiapine Monotherapy in Ambulatory Bipolar Spectrum Disorder With Moderate-to-Severe Hypomanic Symptoms or Mild Manic Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: AstraZeneca (Industry); University of Cincinnati (Other)
Responsible Party: Susan L. McElroy, MD/Professor, Lindner Center of HOPE
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRUSQUET0302
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Bipolar Disorder
Keywords: currently experiencing hypomania or mild mania
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: Quetiapine — Oral dosing: 50mg (Day 1), 100mg (Day 2), 150mg (Day 3), 200mg (Day 4), followed by flexible dosing from 50mg to 800mg through day 56.

SUMMARY:
The purpose of this research study is to evaluate the safety, tolerability, and efficacy of quetiapine compared to placebo (sugar pill without medication) in the treatment of bipolar disorder with moderate to severe hypomania or mild mania. Quetiapine is approved by the United States Food and Drug Administration (FDA) for the treatment of schizophrenia and bipolar mania.

DETAILED DESCRIPTION:
Methods and Procedures

This is a single center, eight-week, randomized, double-blind, placebo-controlled, parallel group, flexible-dose study in 40 outpatients with bipolar disorder types I, II, or NOS by DSM-IV-TR criteria who also have moderate-to-severe hypomanic symptoms or mild manic symptoms (defined as a score of > 3 but <5 on the Clinical Global Impressions Scale Modified for Bipolar Disorder [CGI-BP]). Subjects may have concurrent depressive or anxiety symptoms or syndromes, but they may not have psychotic features (as defined in DSM-IV) or substance dependence. The primary outcome measure will be change in the Young Mania Rating Scale (YMRS) scores. Secondary outcome measures will include the total of the YMRS and the Inventory for Depressive Symptoms (IDS), the IDS alone, the Hamilton Rating Scale for Anxiety (HAM-A), the CGI-BP, the Global Assessment of Functioning (GAF), the Life Functioning Questionnaire (LFQ), and the Sheehan Disability Scale (DSD). Of note, the YMRS-IDS total reflects a novel means of assessing total affective burden. Also, IDS will be used to assess depressive symptoms because of our experience in the Stanley Foundation Bipolar Network indicating that this scale better assesses the signs and symptoms of bipolar depression as compared to both the Hamilton Rating Scale for Depression (HAM-D) and the Montgomery-Asberg Depression Scale (MADRAS). The LFQ is a validated gender neutral scale specifically designed to assess functional outcome in bipolar disorder. The Abnormal Involuntary Movement Scale (AIMS), Simpson Angus Scale (SAS), and Barnes Akathisia Scale (BARS), will be used to assess for degree and severity of extrapyramidal side effects experienced.

Data Analysis and Data Monitoring

All subjects with observations available from the baseline and at least one post-baseline visit will be included in analyses. The primary outcome measure will be the change in YMRS scale scores from baseline to last observation. The difference in YMRS change between treatment groups will be tested for significance (alpha=0.05, two-tailed) using an independent-samples t-test. Measures of change in total affective burden, depressive and anxiety symptoms, global improvement, use of adjunctive anxiolytic and hypnotic medication, adherence to study medication, frequency and severity of side effects, and reasons for early termination will also be analyzed. The final dose achieved by each subject will be correlated with scale score change. Tolerability will be assessed based on adverse experiences, clinical laboratory tests, vital signs (blood pressure and pulse), weight, and discontinuation rates.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years of age or older.
2. Subjects must have bipolar I, II, or not otherwise specified (NOS) disorder as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria. Of note, bipolar NOS disorder will include subjects with either recurrent or sporadic brief hypomanias (hypomanias of 1 to 3 days in duration).
3. Subjects must have moderate-to-severe hypomanic symptoms or mild manic symptoms that must be clinically significant (at least mild) but no worse than moderately severe, defined as a CGI-BP scale for mania > 3 and < 5, on at least 2 assessment days at least 3 days apart during the screening phase.
4. Subjects must not be receiving mood stabilizing, antidepressant, or antipsychotic medication for > one week.
5. Subjects or their legally authorized representative must sign the Informed Consent document after the nature of the trial has been fully explained.
6. If female, subjects must be: postmenopausal, surgically incapable of childbearing, or practicing medically acceptable, effective method(s) of contraception (e.g., hormonal methods, intrauterine device) for at least one month prior to study entry and throughout the study.

Exclusion Criteria:

Criteria for exclusion from this study will be any of the following:

1. Subjects who do not have bipolar disorder by DSM-IV-TR criteria.
2. Subjects who are receiving treatment with an antimanic or mood stabilizing medication (lithium, valproate, carbamazepine, or an antipsychotic), and in the investigators' judgment, require ongoing treatment with that medication.
3. Subjects whose bipolar manic symptoms are presently less than mild (CGI-BP < 2) or more than markedly ill (CGI-BP > 5 or YMRS > 21)
4. Subjects who have severe depressive symptoms (IDS > 39 ) or psychotic features (as defined in DSM-IV)
5. Subjects with clinically significant suicidal or homicidal ideation.
6. Subjects with a current DSM-IV Axis I diagnosis of delirium, dementia, amnesia, or other cognitive disorders; a DSM-IV diagnosis of a substance use disorder within the past six months; a lifetime DSM-IV psychotic disorder (e.g., schizophrenia or schizoaffective disorder).
7. Subjects with serious general medical illnesses including hepatic, renal, respiratory, cardiovascular, endocrine, neurologic, or hematologic disease as determined by the clinical judgment of the clinical investigator. Subjects with hypo- or hyperthyroidism unless stabilized on thyroid replacement > 3 months.
8. Subjects who are allergic to or who have demonstrated hypersensitivity to quetiapine.
9. Women who are pregnant or nursing.
10. Subjects who have received an experimental drug or used an experimental device within 30 days.
11. Subjects who have a history of neuroleptic malignant syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change in manic symptoms (as measured by Young Mania Rating Scale) | baseline to endpoint

SECONDARY OUTCOMES:
Change in total burden of affective symptoms, depressive symptoms alone, and anxiety symptoms alone; change in clinical global improvement; adherence with study medication; and degree and severity of side effects experienced. | baseline to endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Susan L. McElroy, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] McElroy SL, Martens BE, Winstanley EL, Creech R, Malhotra S, Keck PE Jr. Placebo-controlled study of quetiapine monotherapy in ambulatory bipolar spectrum disorder with moderate-to-severe hypomania or mild mania. J Affect Disord. 2010 Jul;124(1-2):157-63. doi: 10.1016/j.jad.2009.11.014. Epub 2009 Dec 5. PMID 19963274